CLINICAL TRIAL: NCT04693858
Title: Enhancing the Capacity of School Nurses to Reduce Excessive Anxiety in Children: an Efficacy Trial of the CALM Intervention
Brief Title: Efficacy Trial of the CALM Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Golda S. Ginsburg, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-037-2; R305A200195 (Other Grant/Funding Number: Institute of Education Sciences)
Record Dates: First submitted 2020-12-14; First posted 2021-01-05 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Anxiety Disorder of Childhood
Keywords: Anxiety; Child anxiety; School-based interventions; School nursing; Brief anxiety interventions; Cognitive-behavioral therapy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study involves a cluster-randomized controlled trial to compare CALM to CALM-R and a weighted waitlist control (WLC) group (4 CALM/CALM-R:1 WLC).
Who Masked: Outcomes Assessor
Masking Description: The Independent Evaluators (IEs) responsible for baseline, post-intervention, and follow-up outcomes assessment will be masked to intervention conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Child Anxiety Learning Modules (CALM) (Experimental): Children randomly assigned to this condition will receive the CALM intervention.
  Interventions: Behavioral: Child Anxiety Learning Modules (CALM)
- Child Anxiety Learning Modules--Relaxation (CALM-R) (Active Comparator): Children randomly assigned to this condition will receive the CALM-R intervention.
  Interventions: Behavioral: Child Anxiety Learning Modules--Relaxation (CALM-R)
- Waitlist control (No Intervention): Within each nurse, 20% (1 in 5) children will be randomly assigned to wait a period of eight weeks prior to starting the intervention with their school nurse. During this period, the child is not prevented from seeing the school nurse, nor are they prevented from continuing to utilize stable doses of community treatment (i.e., therapy outside of school or medication); nurses are simply asked to provide normal support and avoid using techniques specific to CALM or CALM-R. After the 8 weeks, youth are re-evaluated and nurses begin delivering the intervention to the student.

INTERVENTIONS:
Behavioral: Child Anxiety Learning Modules (CALM) — CALM is a cognitive-behavioral intervention for childhood anxiety. CALM consists of five modules. The primary components include psychoeducation, relaxation training (C), behavioral exposure (A), cognitive restructuring (L), and relapse prevention (M). There is also an optional parent psychoeducation module. Students randomized to the CALM condition will receive the 5 modules over 8 weeks.
  Arms: Child Anxiety Learning Modules (CALM)
Behavioral: Child Anxiety Learning Modules--Relaxation (CALM-R) — CALM-R serves as an active comparison condition to CALM and consists of 5 modules of relaxation skills. The key components of CALM-R include psychoeducation, deep breathing, progressive muscle relaxation, guided imagery, and relapse prevention. Students randomized to the CALM-R condition will receive the 5 modules over 8 weeks.
  Arms: Child Anxiety Learning Modules--Relaxation (CALM-R)

SUMMARY:
Excessive anxiety among elementary students is highly prevalent and associated with impairment in academic, social, and behavioral functioning. The primary aim of this project is to evaluate the initial efficacy of a brief nurse-delivered intervention (CALM: Child Anxiety Learning Modules), relative to a credible comparison (CALM-R, relaxation skills only) and a waitlist control for reducing anxiety symptoms and improving education outcomes at post intervention and at a 1-year follow-up. In addition, the research team will assess the cost effectiveness of CALM versus CALM-R and the waitlist control and examine potential predictors, moderators, and mediators of CALM's impact on child outcomes based on the proposed theory of change.

DETAILED DESCRIPTION:
Excessive anxiety among elementary age students is common, severely impairs academic, social, and behavioral functioning, and is associated with significant educational and health care costs. Despite the high burden of anxiety, less than half of children with anxiety receive the services they need to succeed in school. School clinicians can and do support these youth, however, their caseloads are high and their time to provide individualized services is limited. Consequently, there is a critical need to expand the network of providers who can assist students with anxiety and address this malleable obstacle to student academic success. Because somatic complaints, such as headaches and stomach aches, are a hallmark feature of excessive anxiety, school nurses are often the first school-based personnel to identify problematic anxiety in students. However, school nurses currently lack training in evidenced-based anxiety reduction interventions. The current study leverages findings from a three-year IES Development award (R305A140694), through which our team developed and assessed the feasibility of training elementary school nurses to use a brief intervention to reduce student anxiety; it was demonstrated that the training and intervention (i.e., Child Anxiety Learning Modules; CALM) was indeed feasible to implement and resulted in positive changes in student outcomes. CALM is now a fully developed intervention with ready-to-use intervention components and materials, training and coaching procedures, and is ready for an initial efficacy evaluation in authentic school settings. Toward that end, the primary purpose of this study is to evaluate the efficacy of CALM in a fully powered randomized controlled trial. CALM will be delivered by elementary school nurses in rural, suburban, and urban elementary schools nationwide to enhance the generalizability of findings across socioeconomic, racial, ethnic, and neighborhood settings (as approximately 80% of schools in the US have a school nurse). The efficacy of CALM will be tested using gold standard methods (e.g., independent evaluators to assess primary outcomes). The study's primary aim is to evaluate the efficacy of CALM, compared to a credible comparison condition (CALM-R; a school nurse delivered relaxation skills only intervention that parallels CALM in time and format) as well as a waitlist control, for reducing anxiety symptoms and improving educational outcomes at post-intervention and a one year follow-up. The secondary aim is to examine the cost effectiveness of CALM relative to CALM-R and the waitlist control. An exploratory aim is to examine potential predictors, moderators, and mediators of student outcomes based on the proposed theory of change. If efficacious, CALM will be the first evidenced-based school nurse delivered intervention to assist youth with excessive anxiety, filling an important gap in current practices.

ELIGIBILITY:
Student Inclusion Criteria:

* Be between the ages of 5-12
* Have elevated anxiety symptoms as indicated by a) a total SCARED score of 15 or higher based on parent and/or child report using the full SCARED from the baseline evaluation, and/or b) a Clinician Severity Rating of 3 or higher on any anxiety diagnosis from the Anxiety Disorders Interview Schedule for Children DSM-V (ADIS)
* Be fluent in English in order to provide informed consent and assent for their participation and to complete the study measures.
* Children on a stable dose of pharmacological/psychotherapeutic treatment will be eligible as long as the dose has been stable for at least 4 weeks and no changes are considered for the duration of the intervention phase of the study (8 weeks)

Student Exclusion Criteria:

* Children who do not meet the inclusion criteria

Nurse Inclusion Criteria:

* Nurses must be a Registered Nurse (RN) or another similar medical professional
* Nurses must be work in the role of a school nurse
* Nurses must be fluent in English

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 218 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2026-07-03 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression - Impairment (CGI-I) Scale, 8 weeks after baseline | 8 weeks after baseline
  The CGI-I provides a global rating of improvement in anxiety, relative to baseline. The measure yields a single rating of clinical improvement during the past week, relative to the baseline rating. Scores range from 1 (very much improved) to 7 (very much worse).
Clinical Global Impression - Impairment (CGI-I) Scale, 12-month follow-up | 12-month follow-up
  The CGI-I provides a global rating of improvement in anxiety, relative to baseline. The measure yields a single rating of clinical improvement during the past week, relative to the baseline rating. Scores range from 1 (very much improved) to 7 (very much worse).

SECONDARY OUTCOMES:
Children's Somatization Inventory (CSI-24) | Baseline, 8 weeks after baseline, 12-month follow-up
  The CSI-24 is a is 24-item child- and parent-report measure of the child's somatic symptoms. Parents and children respond to the items using a 5-point scale ranging from "not at all" to "a whole lot." One total score calculated by summing the items. Items are scored 0-4 (range: 0-96); higher scores reflect higher levels of subjective severity of somatic symptoms.
Behavioral Avoidance | Baseline, 8 weeks after baseline, 12-month follow-up
  The Behavioral Avoidance form is a 3-item measure assesses how frequently the student avoids specific anxiety provoking situations. The independent evaluator creates a list of the top 3 anxiety-provoking situations and estimates the frequency with which the child avoids those situations over a two week period prior to evaluation. Avoidance for each situation is measured on a 7-point Likert scale, ranging from 1 (never avoid) to 7 (avoid every time).
Children's Automatic Thoughts Scale (CATS) | Baseline, 8 weeks after baseline, 12-month follow-up
  The CATS is a 40-item measure that assesses frequency of students' maladaptive thoughts associated with anxiety. Children respond to items using a 5-point Likert-type scale describing the frequency with which they have had various thoughts over the past week (not at all, sometimes, fairly often, often, all the time). Higher scores reflect greater frequency of negative self-statements. Three scores are derived from the CATS: one total score (20 items, score range 0-80) plus two subscale scores reflecting the content of self-statements: physical threat (10 items, score range 0-40), social threat (10 items, score range 0-40).
Children's Global Assessment Scale (CGAS) | Baseline, 8 weeks after baseline, 12-month follow-up
  The CGAS is a rating scale that indicates a child's global functioning on a scale of 1 (lowest) to 100 (highest). In general, scores below 70 are indicative of increasingly severe impairment in functioning.
Student Attendance Form | Two weeks prior to the evaluations
  The student attendance form is completed by teachers to assess the child's recent (past two weeks) school attendance including number of full and partial days missed as well as the amount of extra time and attention spent on the child.
School Attendance and Discipline | Baseline, 8 weeks after baseline, 12-month follow-up
  The School Attendance and Discipline form is an 8-item measure completed by parents that collects information regarding absences from school related to emotional/behavioral problems as well as disciplinary actions at school.
Student school records - attendance | Baseline, 8 weeks after baseline, 12-month follow-up
  Student records will be obtained from the school that will provide information regarding number of absences, tardiness, and early dismissals during the marking period closest to the dates of baseline, 8-weeks after baseline, and 12-month follow up
Student school records - disciplinary actions | Baseline, 8 weeks after baseline, 12-month follow-up
  Student records will be obtained from the school that will provide information regarding number of referrals for disciplinary action during the marking period closest to the dates of baseline, 8-weeks after baseline, and 12-month follow up
Student school records - grades | Baseline, 8 weeks after baseline, 12-month follow-up
  Student records will be obtained from the school that will provide information regarding English and math grades, as well as any grade retention during the marking period closest to the dates of baseline, 8-weeks after baseline, and 12-month follow up. Grades will be categorized into 4 categories: below expectations/not meeting expectations/needs more time (D); near expectations/exhibits progress towards meeting expectations/developing (C); meets expectations/consistently evident (B); exceeds expectations (A)
Student school records - special education | Baseline, 8 weeks after baseline, 12-month follow-up
  Student records will be obtained from the school that will provide information regarding if the student received special education services (i.e., 504 plan and/or IEP) during the marking period closest to the dates of baseline, 8-weeks after baseline, and 12-month follow up
Subtests from the Woodcock-Johnson Tests -Achievement and Cognitive Batteries (WJ IV) | Baseline, 8 weeks after baseline, 12-month follow-up
  Subtests from the WJ-IV (i.e., reading, math fluency, and digits backwards) will be administered by the IE to measure cognitive factors (e.g., efficiency, speed, working memory) that are believed to be affected by anxiety. Standard scores will be derived for the Reading Sentences Fluency, Math Facts Fluency, and Numbers Reversed subtests. Standard scores reflect the following ability level: <69=very low; 70-79=low; 80-89=low average; 90-110=average; 111-120=high average; 121-130=superior; >131=very superior.
Strength and Difficulties Questionnaire (SDQ), Teacher and Parent Versions | Baseline, 8 weeks after baseline, 12-month follow-up
  The SDQ assesses a range of emotional and behavioral difficulties in children 4-17 years old (e.g., conduct problems, hyperactivity/ inattention, peer relationship problems, and prosocial behaviors). Nine scores can be derived from the SDQ. (1-5) Five subscales, each of which corresponds to 5 domains: emotional symptoms, conduct problems, hyperactivity, peer problems, prosocial problems. Subscale scores are summed. (6) The total score is generated by summing the scores from all the scales except the prosocial scale. (7-8) Externalizing scores (conduct and hyperactivity) and internalizing scores (emotional and peer problems) are also provided. (9) The impact score is a sum of questions reflecting distress and impairment. Subscale scores each range from 0-10. Externalizing and internalizing scores range from 0-20. The total score can range from 0 to 40. The impact score ranges from 0-6. Higher scores indicate higher levels of the behavior in question.
Teacher Observation of Classroom Adaptation-Checklist Concentration subscale (TOCA-C) | Baseline, 8 weeks after baseline, 12-month follow-up
  The TOCA-C concentration subscale is a 7-item subscale of the TOCA that assesses teachers' perceptions of a student's classroom concentration problems. Teachers rate student concentration on a 6-point Likert scale that ranges from "never (1)" to "almost always (6)." Only the Concentration Problems subscale is used in this study. This subscale includes 7 items (range = 7-42). Higher scores on indicate more maladaptive behaviors.
Academic Competence Evaluation Scale (ACES), short version | Baseline, 8 weeks after baseline, 12-month follow-up
  The ACES is a 32-item teacher report measure that assesses classroom skills and behaviors. Each item is rated on a 5 point scale (1 = never, 5= almost always), with the option to indicate that the behavior is not observed (N/O). The measure is divided in 2 main scales: Academic Skills (14, score range 0-70), consisting of Reading/Language Arts (6 items, score range 0-30), Mathematics (4 items, score range 0-20), and Critical Thinking (4 items, score range 0-20); Academic Enablers (18 items, score range 0-90), consisting of Motivation (5 items, score range 0-25), Engagement (4 items, score range 0-20), Study Skills (4 items, score range 0-20), and Interpersonal Skills (5 items, score range 0-25). Higher scores reflect higher abilities.
Child Anxiety Impact Scale (CAIS) | Baseline, 8 weeks after baseline, 12-month follow-up
  The CAIS is a 27-item child- and parent-report measure of anxiety-related interference in social, academic and family functioning. Children and parents respond to items using a 4-point Likert scale (not at all, just a little, pretty much, very much); higher scores represent greater interference of anxiety in child functioning. The CAIS-C has a total score (27 items, score range 0-81) and three subscales: school (10 items, score range 0-30), social (11 items, score range 0-33), and home/family (6 items, score range 0-18).
School Anxiety Scale - Teacher Report (SAS-TR) | Baseline, 8 weeks after baseline, 12-month follow-up
  The SAS is a 16-item teacher questionnaire that assesses anxiety in the school setting, with a specific focus on social and generalized anxiety symptoms relevant to classroom participation. Teachers rate student anxiety on a 4-point Likert scale that ranges from "never (0)" to "always (3)." The SAS-TR contains a total score (16 items, range of 0 to 48) and two subscales: social anxiety (7 items, range of 0-21) and generalized anxiety (9 items, range of 0 to 27). Higher scores represent higher levels of anxiety; scores of 8 and more on the social anxiety, 10 or more on the generalized anxiety, and 17 or more on the total anxiety is considered to represent high anxious condition.
Clinical Global Impression - Severity (CGI-S) Scale | Baseline, 8 weeks after baseline, 12-month follow-up
  The CGI-S provides a global rating of anxiety severity. The measure yields a single rating of anxiety symptom severity during the past week. Scores range from 1 (Normal; Not at all ill) to 7 (Extremely ill)
Anxiety Disorders Interview Schedule for DSM-V, Parent and Child Versions (ADIS-V) | Baseline, 8 weeks after baseline, 12-month follow-up
  The ADIS-V is a structured interview that assesses anxiety diagnoses and severity in youth. Impairment ratings are generated for each diagnosis using the Clinician Severity Rating (CSR, range = 0-8; higher CSRs indicate higher severity of anxiety disorders, a CSR of 4 is required to assign a diagnosis). Diagnoses are derived separately from the child and parent report, which yields a Composite Diagnosis that is one measure used to determine study eligibility.
Screen for Child Anxiety-Related Emotional Disorders (SCARED), parent and child versions | Baseline, 8 weeks after baseline, 12-month follow-up
  The SCARED is a 41-item child- and parent-report measure of anxiety. Youth and parents respond to items using a 3-point Likert-type scale describing the degree to which statements are true (0 = not true or hardly ever true, 1 = somewhat true or sometimes true, 2 = very true or often true). Higher scores represent higher levels of anxiety. Six scores can be derived from the SCARED: one total score (41 items, score range 0-82) plus five subscale scores: panic/somatic (13 items, score range 0-26), generalized anxiety (9 items, score range 0-18), (3) separation anxiety (8 items, score range 0-16), social anxiety (7 items, score range 0-14), and school phobia (4 items, score range 0-8).

OTHER OUTCOMES:
CALM and CALM-R Intervention Fidelity, Adherence, Differentiation, and Competence | After each session of the CALM or CALM-R intervention is delivered (approximately 1 session of the intervention delivered each week, for up to 8 weeks)
  The CALM and CALM-R Intervention Fidelity, Adherence, Differentiation, and Competence forms contain key points/principles that should be covered during each CALM and CALM-R module and assesses whether they were covered (yes/no), the quality of administration (using a 4 point scale where 1 = poor to 4 = very good), and non-specific factors (e. g., maintains a positive working relationship). For adherence, a yes indicates nurses adhere to the manual; no indicates nurses did not adhere for that particular item. For quality, highest scores indicate greater quality of competence in delivering the intervention components.
Independent Evaluator (IE) masking form | After post (8-week) and follow up (12-month) evaluations
  The IE masking form is a 1-item measure that asks the IE to guess the student's intervention assignment in order to assess the integrity of the masking procedures.
Session Summary Form (SSF) | After each session of the CALM or CALM-R intervention is delivered (approximately 1 session of the intervention delivered each week, for up to 8 weeks)
  The SSF captures pertinent information about the session such as duration, attendance, intervention strategy, and ratings of the quality of the therapeutic relationship, child compliance, and nurse's perceived competence.
Nurse Background Form | Baseline
  The nurse background form assesses demographic characteristics and professional experience (e.g., training, years of experience, license).
Maslach Burnout Inventory - General Survey | Baseline, 8 weeks after baseline (with each child), 12-month follow-up
  The Maslach Burnout Inventory - General Survey is a 16-item measure completed by nurses that assesses overall levels of burnout on a 6-point likert scale (0=never, 6=every day; scores range from 0-96), with higher scores indicating higher levels of burnout. There are three subscales: exhaustion (5 items, score range 0-30), cynicism (5 items, score range 0-30), and personal efficacy (reverse-scored; 6 items, score range 0-36)
Student-Nurse Relationship Scale -Closeness Subscales, student and nurse reports | Baseline, 8 weeks after baseline
  The student-nurse relationship scale is a 7-item assesses the quality of the student-nurse relationship on a _-point Likert scale (1=definitely does not apply/is not true, 5=definitely applies/is true); scores range from 7-35), with higher scores indicating a stronger relationship.
Family demographic form | Baseline
  The family demographic form collects information from the parent about the child and the family including age, sex, race, economic status, household family members and parents' marital status.
Willingness-to-Pay (WTP) questionnaire | At the conclusion of the CALM study (4 years following the beginning of the study)
  The WTP questionnaire obtains a dollar-denominated measure of CALM sites' principals/senior administrator willingness to support the implementation of CALM in their schools and therefore to re-allocate a portion of their budgets to the costs of implementing, operating, and sustaining CALM.
Child Health Utility 9-D Index (CHUD) | Baseline, 8 weeks after baseline, 12-month follow-up
  The CHUD is a population-based preference-weighted utility index for use in cost-effectiveness analyses. There are a total of 9 dimensions/items (worried, sad, pain, tired, annoyed, schoolwork/homework, sleep, daily routine, and joining in activities) with 5 levels within each dimension. Parents are asked to indicate which level within each dimension is most like their child on the day that they complete the questionnaire. Scores range between 0.33 and 1. Higher scores reflect poorer overall general health-related quality of life.
Child and Adolescent Services Assessment (CASA) | Baseline, 8 weeks after baseline, 12-month follow-up
  The CASA is a 20-item measure that assesses use of general medical health, mental health, social service, and education services. Items are dichotomous (no=0, yes=1), with checkboxes to indicate details about services (e.g., frequency, indication, provider).
Parent's missed work form | Baseline, 8 weeks after baseline, 12-month follow-up
  This form asks parents to report their total missed days of work due to emotional difficulties of their child.
Nurse time logs | Baseline, weekly, 8 weeks after baseline, 12-month follow-up
  Nurses will complete time logs for each encounter with students enrolled in the study; these logs are used to capture the amount of time spent by the school nurse addressing the needs of the anxious child - at any time - during the active intervention phase (from enrollment through last session). Nurses will record the start and end times of each encounter and a brief checklist of intervention tasks completed, and will also record any other tasks they completed in connection with the encounters, including any communication with school staff members or parents.

CONTACTS AND LOCATIONS:
Overall Officials: Golda S Ginsburg, Ph.D., Principal Investigator — UConn Health; Kelly Drake, Ph.D., Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - University of Connecticut School of Medicine, West Hartford, Connecticut
  - Anxiety Treatment Center of Maryland, Columbia, Maryland

IPD SHARING:
Plan to Share IPD: Yes
1. Publications: we will submit all publications to the ERIC within 12 months of the publisher's official date of final publication. We will also email copies of publications to interested parties upon request.
  2. Data Access/Sharing: We will provide timely access to the final research data (including data file in SPSS format and a variable codebook). We will share only cleaned, de-identified or synthetic data. These data include surveys/interviews and school records. We will create a data documentation file (i.e., description of all original and derived/summary variables and definitions) to accompany the data file. The documentation will include a description of the study, data collection forms, study protocol/procedures, descriptions of variable recoding performed, and a list of major study publications and investigators.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The de-identified data and documentation files will be available after the final wave of data are collected, cleaned, and the primary outcome manuscript has been accepted for publication. The data will remain accessible for at least 10 years and the timeframe of data accessibility will be reviewed at the annual progress reviews and revised as necessary.
Access Criteria: A a CALM Data Request Form will be required from interested individuals. Data will be sent under conditions that the request is reasonable and will be provided to qualified researchers or allied professionals with the necessary skills to use and interpret the data responsibly.

REFERENCES:
- [Background] Ginsburg GS, Drake KL, Muggeo MA, Stewart CE, Pikulski PJ, Zheng D, Harel O. A pilot RCT of a school nurse delivered intervention to reduce student anxiety. J Clin Child Adolesc Psychol. 2021 Mar-Apr;50(2):177-186. doi: 10.1080/15374416.2019.1630833. Epub 2019 Aug 2. PMID 31373524
- [Background] Drake KL, Stewart CE, Muggeo MA, Ginsburg GS. Enhancing the Capacity of School Nurses to Reduce Excessive Anxiety in Children: Development of the CALM Intervention. J Child Adolesc Psychiatr Nurs. 2015 Aug;28(3):121-30. doi: 10.1111/jcap.12115. Epub 2015 Jul 14. PMID 26171792
- [Background] Muggeo, M. A., Stewart, C. E., Drake, K. L., & Ginsburg, G. S. (2017). A school nurse-delivered intervention for anxious children: An open trial. School Mental Health, 9(2) 157-171.